CLINICAL TRIAL: NCT01245374
Title: Assessment of the Ease of Use of Norditropin NordiFlex® Relative to the One of the Device Previously Used by Patients or Parents
Brief Title: Norditropin NordiFlex® Device Compared to the Device Previously Used by Patients or Parents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GH-3826; U1111-1117-1194 (Other: WHO); 2009-017387-16 (EudraCT Number)
Record Dates: First submitted 2010-11-19; First posted 2010-11-22 (Estimated); Results first posted 2012-06-25 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-01

CONDITIONS: Growth Hormone Disorder; Growth Hormone Deficiency in Children; Foetal Growth Problem; Small for Gestational Age; Genetic Disorder; Turner Syndrome; Chronic Kidney Disease; Chronic Renal Insufficiency; Delivery Systems
MeSH Terms: conditions — Genetic Diseases, Inborn; Turner Syndrome; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nordiflex Norditropin® (Experimental): Individually adjusted dose administered with Norditropin NordiFlex® for 6 weeks. Dosage depended on age, weight, etiologies and according to the summary of product characteristics (SPC)
  Interventions: Device: Norditropin NordiFlex®

INTERVENTIONS:
Device: Norditropin NordiFlex® — Daily administration by a subcutaneous injection (under the skin). Starting dose and frequency will be determined by the physician as part of normal clinical practice

SUMMARY:
This study is conducted in Europe. The aim of this study is to compare the easiness of use of Norditropin NordiFlex® device to the device previously used by patients or parents.

ELIGIBILITY:
Inclusion Criteria:

* Children who can receive Norditropin® (somatropin) treatment according to the product labelling
* Treated with growth hormone for at least one year

Exclusion Criteria:

* Contraindications to Norditropin® growth hormone therapy
* Known or suspected hypersensitivity to somatropin or related products
* The receipt of any investigational medicinal product within 3 months prior to study start
* Life threatening disease, for example cancer
* Pregnancy or the intention of becoming pregnant

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2010-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Paris La Défense Cedex, France

REFERENCES:
- [Result] Tauber M, Jaquet D, Jesuran-Perelroizen M, Petrus M, Bertrand AM, Coutant R; NordiFlex(R) French Study Group. User assessment of Norditropin NordiFlex((R)), a new prefilled growth hormone pen: a Phase IV multicenter prospective study. Patient Prefer Adherence. 2013 May 24;7:455-62. doi: 10.2147/PPA.S43460. Print 2013. PMID 23737664
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted in France (38 sites). Recruitment period occurred from 17-Nov-2010 to 18-Apr-2011.
Pre-assignment Details: Eligible participants had to receive training for the use of Nordiflex® system. A member of the investigator's team, physician or nurse, was in charge of this training. At inclusion and before receiving treatment, participants or parents had to complete a questionnaire about the ease of use of the previously used device.
Groups:
- Norditropin NordiFlex®: Individually adjusted dose administered with Norditropin NordiFlex® for 6 weeks. Dosage depended on age, weight, etiologies and according to the summary of product characteristics (SPC).
Period: Overall Study
Arm/Group | Norditropin NordiFlex®
Started | 103
Completed | 99
Not Completed | 4
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Norditropin NordiFlex®
Number analyzed (Participants) | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.7 (2.94)
Gender [Count of Participants; unit: Participants]
  Female | 43
  Male | 60
Region of Enrollment [Number; unit: participants]
  France | 103
Height [Mean (Standard Deviation); unit: cm] | 141.0 (16.5)
Weight [Mean (Standard Deviation); unit: kg] | 37.3 (16.0)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 18.1 (4.26)
Duration of growth hormone treatment [Mean (Standard Deviation); unit: years] | 4.18 (2.81)

OUTCOME MEASURES:

1. Primary Outcome: The Relative Ease of Use of NordiFlex® Compared to the Device Previously Used
Description: Analysed for the ITT (intent-to-treat) analysis set: The relative ease of use of the trial injection device compared to the device previously used was assessed using a quantitative scale, ranging from 0 to 10 with 0 = NordiFlex® is far less simple, 5 = equivalent simplicity and 10 = NordiFlex® is far more simple. The participants had to circle the number that represented their perception of the current state.
Time Frame: Week 6
Population: Intent-to-treat (ITT) consists of all participants included in the trial and having signed the informed consent form.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Norditropin NordiFlex®
Number analyzed (Participants) | 103
units on a scale | 6.89 (2.52)

2. Primary Outcome: The Relative Ease of Use of NordiFlex® Compared to the Device Previously Used
Description: Analysed for the PP (per protocol) analysis set: The relative ease of use of the trial injection device compared to the device previously used was assessed using a quantitative scale, ranging from 0 to 10 with 0 = NordiFlex® is far less simple, 5 = equivalent simplicity and 10 = NordiFlex® is far more simple. The participants had to circle the number that represented their perception of the current state.
Time Frame: Week 6
Population: Per protocol set (PP): All subjects in the ITT set using NordiFlex® and had completed the trial without any significant violation of the inclusion/exclusion criteria or any other aspect of the protocol considered to potentially affect the efficacy results.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Norditropin NordiFlex®
Number analyzed (Participants) | 98
units on a scale | 6.98 (2.46)

3. Secondary Outcome: Percentage of Participants Evaluating Simplicity of Use: Dose Selection Easiness
Description: The overall simplicity of use was evaluated at every step of the injection preparation (dose selection, injection and dose modification) and using the time spent in the preparation of the injection. Ordinal variables were used for the evaluation (very easy, easy, fairly easy, difficult and very difficult).
Time Frame: Week 0
Population: Intent-to-treat (ITT) consists of all participants included in the trial and having signed the informed consent form.
Measure: Number; unit: percentage of participants
Arm/Group | Norditropin NordiFlex®
Number analyzed (Participants) | 103
percentage of participants
  Very easy | 55.3
  Easy | 38.8
  Fairly easy | 4.85
  Difficult | 0.97
  Very difficult | 0

4. Secondary Outcome: Percentage of Participants Evaluating Simplicity of Use: Dose Modification
Description: as for outcome 3
Time Frame: Week 0
Population: Intent-to-treat (ITT) consists of all participants included in the trial and having signed the informed consent form. For seven patients, no data available.
Measure: Number; unit: percentage of participants
Arm/Group | Norditropin NordiFlex®
Number analyzed (Participants) | 96
percentage of participants
  Very easy | 26.0
  Easy | 40.6
  Fairly easy | 19.8
  Difficult | 11.5
  Very difficult | 2.08

5. Secondary Outcome: Percentage of Participants Evaluating Simplicity of Use: Injection Easiness
Description: as for outcome 3
Time Frame: Week 0
Population: Intent-to-treat (ITT) consists of all participants included in the trial and having signed the informed consent form. For three patients, no data available.
Measure: Number; unit: percentage of participants
Arm/Group | Norditropin NordiFlex®
Number analyzed (Participants) | 100
percentage of participants
  Very easy | 44.7
  Easy | 43.7
  Fairly easy | 9.71
  Difficult | 1.94
  Very difficult | 0

6. Secondary Outcome: Percentage of Participants Evaluating Simplicity of Use: Time Spent in the Preparation of the Injection
Description: The overall simplicity of use was evaluated at every step of the injection preparation (dose selection, injection and dose modification) and using the time spent in the preparation of the injection. This was evaluated using time intervals: below 5 minutes, 5-10 minutes, 10-20 minutes.
Time Frame: Week 0
Population: Intent-to-treat (ITT) consists of all participants included in the trial and having signed the informed consent form.
Measure: Number; unit: percentage of participants
Arm/Group | Norditropin NordiFlex®
Number analyzed (Participants) | 103
percentage of participants
  Below 5 minutes | 86.4
  5-10 minutes | 11.7
  10-20 minutes | 1.94

7. Secondary Outcome: Percentage of Participants Evaluating Simplicity of Use: Dose Selection Easiness
Description: as for outcome 3
Time Frame: Week 6
Population: Intent-to-treat (ITT) consists of all participants included in the trial and having signed the informed consent form.
  For one patient, no data available.
Measure: Number; unit: percentage of participants
Arm/Group | Norditropin NordiFlex®
Number analyzed (Participants) | 102
percentage of participants
  Very easy | 66.7
  Easy | 21.6
  Fairly easy | 8.82
  Difficult | 2.94
  Very difficult | 0

8. Secondary Outcome: Percentage of Participants Evaluating Simplicity of Use: Dose Modification
Description: as for outcome 3
Time Frame: Week 6
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Norditropin NordiFlex®
Number analyzed (Participants) | 100
percentage of participants
  Very easy | 84.0
  Easy | 13.0
  Fairly easy | 2.0
  Difficult | 1.0
  Very difficult | 0.00

9. Secondary Outcome: Percentage of Participants Evaluating Simplicity of Use: Injection Easiness
Description: as for outcome 3
Time Frame: Week 6
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Norditropin NordiFlex®
Number analyzed (Participants) | 102
percentage of participants
  Very easy | 62.7
  Easy | 22.5
  Fairly easy | 12.7
  Difficult | 0.98
  Very difficult | 0.98

10. Secondary Outcome: Percentage of Participants Evaluating Simplicity of Use: Time Spent in the Preparation of the Injection
Description: as for outcome 6
Time Frame: Week 6
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Norditropin NordiFlex®
Number analyzed (Participants) | 102
percentage of participants
  Below 5 minutes | 93.1
  5-10 minutes | 5.88
  10-20 minutes | 0.98

11. Secondary Outcome: Ease of Learning Assessed by the Physician or the Nurse: Ease of Training
Description: The person in charge, physician or nurse, of giving all the instruction of use to patients or parents assessed the ease of learning of the Nordiflex® device. Ease of learning was evaluated using ordinal variables (very easy, easy and difficult).
Time Frame: Week 6
Population: Intent-to-treat (ITT) consists of all participants included in the trial and having signed the informed consent form.
Measure: Number; unit: percentage of participants
Arm/Group | Norditropin NordiFlex®
Number analyzed (Participants) | 103
percentage of participants
  Very easy | 72.8
  Easy | 26.2
  Difficult | 0.97

12. Secondary Outcome: Ease of Learning Assessed by the Physician or the Nurse: Time Learning
Description: The person in charge, physician or nurse, of giving all the instruction of use to patients or parents assessed the ease of learning of the Nordiflex® device. Time to learning was assessed using time intervals: 6-10 minutes, 11-15 minutes, 16-30 minutes and 31 minutes to 1 hour.
Time Frame: Week 6
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Norditropin NordiFlex®
Number analyzed (Participants) | 100
percentage of participants
  6-10 minutes | 40.0
  11-15 minutes | 26.0
  16-30 minutes | 30.0
  31 minutes - 1 hour | 4.0

13. Secondary Outcome: Ease of Learning Assessed by the Physician or the Nurse: Added Values of the Products
Description: The person in charge, physician or nurse, of giving all the instruction of use to patients or parents assessed the ease of learning of the Nordiflex® device. An added value of device was evaluated by the physician or the nurse using categorical variables.
Time Frame: Week 6
Population: Intent-to-treat (ITT) consists of all participants included in the trial and having signed the informed consent form.
Measure: Number; unit: percentage of participants
Arm/Group | Norditropin NordiFlex®
Number analyzed (Participants) | 103
percentage of participants
  Overall simplicity | 82.5
  Dose selection | 35.0
  Maximum available dose | 15.5
  Dose adjustment | 64.1
  Easiness of injection | 26.2
  Improvement of compliance or motivation | 27.2
  No added values | 4.85

14. Secondary Outcome: Patient Autonomy: Percentage of Patients Performing Operations for Treatment Injection
Description: The patient autonomy was evaluated using percentage of participants who performed all the operations of the treatment administration including dose selection, dose modification in case of error and injection.
Time Frame: Week 0
Population: Intent-to-treat (ITT) consists of all participants included in the trial and having signed the informed consent form.
Measure: Number; unit: percentage of participants
Arm/Group | Norditropin NordiFlex®
Number analyzed (Participants) | 103
percentage of participants
  Yes | 28.2
  No | 71.8

15. Secondary Outcome: Patient Autonomy: Percentage of Patients Performing Operations for Treatment Injection
Description: as for outcome 14
Time Frame: Week 6
Population: Intent-to-treat (ITT) consists of all participants included in the trial and having signed the informed consent form.
Measure: Number; unit: percentage of participants
Arm/Group | Norditropin NordiFlex®
Number analyzed (Participants) | 103
percentage of participants
  Yes | 41.2
  No | 58.8

16. Secondary Outcome: Patient Preference: Percentage of Participants Preferring System for Continuation of Growth Hormone Treatment
Description: The patient preference was evaluated using the percentage of participants preferring the new system, old system or none of them for their growth hormone therapy.
Time Frame: Week 6
Population: Intent-to-treat (ITT) consists of all participants included in the trial and having signed the informed consent form. For two patients, no data available.
Measure: Number; unit: percentage of participants
Arm/Group | Norditropin NordiFlex®
Number analyzed (Participants) | 101
percentage of participants
  Nordiflex® | 64.36
  Previous system | 34.65
  None of them | 0.99

17. Secondary Outcome: Number of Participants Reporting Adverse Events, Medical Events of Special Interest (MESI) and Technical Problems With Devices Used in Trial
Time Frame: Weeks 0 - 6
Population: The safety set consisted of all participants included in the trial and having taken at least one dose of trial treatment. The adverse events and technical complaints were collected during the treatment period (6 weeks after inclusion).
Measure: Number; unit: participants
Arm/Group | Norditropin NordiFlex®
Number analyzed (Participants) | 103
participants
  Serious adverse events | 0
  Medical event of special interest (MESI) | 0
  At least one technical complaint | 14
  NordiFlex® pen technical complaint | 8
  PenMate technical complaint | 10
  Other adverse events greater than or equal to 5% | 0

ADVERSE EVENTS:
Time Frame: The adverse events were collected during treatment period (6 weeks after inclusion).
Description: The safety set consisted of all participants included in the trial and having taken at least one dose of trial treatment.
Arm/Group | Norditropin NordiFlex®
Serious Adverse Events (participants affected / at risk) | 0/103
Other Adverse Events (participants affected / at risk) | 0/103

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk reserves the right to not release data until specified milestones, including the right to not release interim results of clinical trials. At the end of the trial, one or more manuscripts for publication will be prepared collaboratively between Investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for less than 60 days to protect intellectual property.